CLINICAL TRIAL: NCT06498934
Title: Deep Brain Stimulation of Cerebellar Dentate Nucleus Promotes Upper Limb Motor Function Recovery After Ischemic Stroke: a Randomized, Double-blind, Sham-controlled Trial
Brief Title: Deep Brain Stimulation of the Dentate Nucleus for Motor Rehabilitation After Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Municipal Administration of Hospitals (Other Government)
Collaborators: Beijing Pins Medical Co., Ltd (Industry)
Responsible Party: Principal Investigator, Zhang Jianguo, Director of functional neurosurgery in Beijing Tiantan Hospital, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HX-A-2024030
Record Dates: First submitted 2024-07-05; First posted 2024-07-12 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Stroke; Upper Extremity Paresis
Keywords: deep brain stimulation; the dentate nucleus
MeSH Terms: conditions — Stroke; Paresis | interventions — Deep Brain Stimulation; Rehabilitation

STUDY DESIGN:
Intervention Model Description: Double blind, randomized, parallel study with partial crossover (control subjects crossover to treatment after randomized portion)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, therapists, care providers, investigators, and outcomes assessors do not know which group (real DN-DBS or control) the patients are randomized. Only the programmer who programs the device settings knows which group the subject is randomized into.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real DN-DBS + rehabilitation (Experimental): Study treatment is deep brain stimulation of the dentate nucleus (DN-DBS) delivered during 6-month rehabilitation period.
  Interventions: Device: deep brain stimulation; Other: Rehabilitation
- sham DN-DBS + rehabilitation (Active Comparator): Active control treatment is rehabilitation (standard-of-care treatment) with sham DN-DBS (electrode implanted but won't turn on the device).
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Device: deep brain stimulation — Stimulation of the dentate nucleus that is paired with upper limb rehabilitation movements.
  Arms: real DN-DBS + rehabilitation
Other: Rehabilitation — Rehabilitation movements to improve upper limb function after stroke

SUMMARY:
The goal of this clinical trial is to learn if deep brain stimulation of the dentate nucleus (DN-DBS) works to promote chronic post-stroke upper limb motor function in adults. It will also learn about the safety of DN-DBS. The main questions it aims to answer are:

Does DN-DBS paired with rehabilitation improve the upper limb motor function of participants more than rehabilitation only? What medical problems do participants have when using DN-DBS for post-stroke rehabilitation?

Researchers will compare real DN-DBS+rehabilitation to sham DN-DBS+rehabilitation (electrodes will be implanted, but no electrical current is given) to see if DN-DBS works to promote chronic post-stroke upper limb motor function.

Participants will:

Undergo unilateral DN-DBS surgery Take real DN-DBS+rehabilitation or sham DN-DBS+rehabilitation as treatment for 6 months Visit the clinic every month during the DN-DBS+rehabilitation (treatment) period for programing, checkups and tests Visit the clinic at Day 1, 30, 90 and 365 after treatment period for checkups and tests

ELIGIBILITY:
Inclusion Criteria:

1. Within the first year to 3 years after the first stroke;
2. Unilateral infarction located in the territory of the middle cerebral artery, but not involving the cerebellum, thalamus, and brainstem;
3. Aged 18-80 years;
4. TMS standard: TMS induces muscle evoked potential (MEP). In the contracted state of the paralyzed muscle (maximum voluntary contraction of 20-50%), a reliable standard MEP (in 5/10 trials with 50-100uv) can be induced;
5. Researchers determine the medical and neurological condition of the participant to be stable based on the participant's medical history, physical examination, and neurological examination;
6. Moderate-severe unilateral upper limb paralysis, i.e., the Fugl-Meyer Assessment (FMA-UE) scale score is ≤47;
7. The distal extremity of the limb has some degree of motor function (flexion of the elbow joint or extension of the elbow joint or partial finger flexion with FMA-UE ≥1);
8. mRS<4 points, able to cooperate with assessment and rehabilitation;
9. No spasticity or mild spasticity in any part of the affected limb (intramuscular rotator muscle and adductor muscle of the shoulder joint, flexor muscle of the elbow joint, flexor muscle of the wrist joint or finger flexor muscle), modified Ashworth scale (MAS) <4 points;
10. MMSE>24 points.

Exclusion Criteria:

1. Primary hemorrhagic stroke or severe hemorrhagic conversion;
2. Any progressive neurological or somatic disease that impairs the function of the affected limb other than stroke;
3. Moderate to severe neglect or disinhibition of the affected limb;
4. Any other neurological disorder that may compromise study safety, including central nervous system vasculitis, intracranial tumors, intracranial aneurysms, multiple sclerosis, or arteriovenous malformations;
5. Pain intensity on the affected limb NRS ≥5 or severe sensory disturbance, NIHSS (item 8) = 2;
6. Exclusion of cardioembolic stroke, patients requiring long-term anticoagulation;
7. Unable to stop anticoagulation treatment at least 10 days prior to surgery (i.e., antiplatelet and/or anticoagulant therapy);
8. Seizure(s) after stroke or potential risk of seizure(s);
9. Switching to oral spasticity medication within 2 weeks of enrollment, or injection of botulinum toxin in the affected arm within 4 months, and/or intention to start taking spasticity medication or inject botulinum toxin during the study follow-up period or within 12 months after implantation;
10. The presence of active psychosis that may affect treatment effect, such as psychosis or severe personality disorder;
11. Untreated or inadequately treated depression, i.e., Beck Depression Inventory score of 20 or more at admission;
12. Diagnosis of dementia;
13. Uncontrolled hypertension or history of cardiovascular disease for a long time;
14. MRI contraindications, such as implanted metal devices or electronic devices (pacemakers, defibrillators, spinal cord stimulators);
15. Participated in another device, biological, or drug study within 30 days of consenting to participate in the current study;
16. Non-pregnant or fertile women must use acceptable contraception, and pregnant women are excluded or terminated from the study;
17. Received decompressive craniectomy;
18. The patient has severe cerebral small vessel disease, basilar artery vascular disease, and/or any other structural abnormalities of the cerebellum, cerebellar peduncles, and brainstem that prevent safe placement of DBS;
19. The investigator determines that the patient has a condition that would significantly increase the risk of study non-compliance, study safety, and/or study integrity. For the safety of the subject, for example, if the subject experiences an exacerbation of their condition, a serious adverse event, or poor compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment, Upper Limb (FMA-UE) Average Change at Day 1 | V6, One day after 6-months of therapy
  The Fugl-Meyer Assessment, Upper Limb (FMA-UE) was analyzed for difference in average change at Day-1 after 6-months of therapy compared to baseline (Difference in average change in FMA-UE from baseline [V0] to one day after therapy [V6]). FMA-UE was collected at each visit. The FMA-UE is a common scale used to measure motor impairment after a stroke. The range is 0 (more impairment) to 66 (no impairment).

SECONDARY OUTCOMES:
Fugl-Meyer Assessment, Upper Limb (FMA-UE) Average Change at Day 90 | V8, 90 days after 6-months of therapy
  The Fugl-Meyer Assessment, Upper Limb (FMA-UE) was analyzed for difference in average change at Day-90 after 6-months of therapy compared to baseline (Difference in average change in FMA-UE from baseline [V0] to 90 days after therapy [V8]). FMA-UE was collected at each visit. The FMA-UE is a common scale used to measure motor impairment after a stroke. The range is 0 (more impairment) to 66 (no impairment).
Wolf Motor Function Test (WMFT) Average Change at Day 1 | V6, One day after 6-months of therapy
  The Wolf Motor Function Test (WMFT) is an assessment scale of upper extremity functional level after stroke. The functional assessment range is an average of 15 sub-items with a range from 0 to 5, with 0 (meaning did not attempt) to 5 (meaning normal). WMFT Day 1 - is a measure of the functional assessment change from baseline to one day after 6-months of therapy.
Wolf Motor Function Test (WMFT) Average Change at Day 90 | V8, 90 days after 6-months of therapy
  The Wolf Motor Function Test (WMFT) is an assessment scale of upper extremity functional level after stroke. The functional assessment range is an average of 15 sub-items with a range from 0 to 5, with 0 (meaning did not attempt) to 5 (meaning normal). WMFT Day 90 - is a measure of the functional assessment change from baseline to 90 days after 6-months of therapy.
Action Research Arm Test (ARAT) Average Change at Day 1 | V6, One day after 6-months of therapy
  Action Research Arm Test (ARAT) is a common scale of fine movements of distal upper limbs after stroke. The functional assessment range is an average of 19 sub-items with a range from 0 to 3, with 0 (meaning did not attempt) to 5 (meaning normal). ARAT Day 1 - is a measure of the functional assessment change from baseline to one day after 6-months of therapy.
Action Research Arm Test (ARAT) Average Change at Day 90 | V8, 90 days after 6-months of therapy
  Action Research Arm Test (ARAT) is a common scale of fine movements of distal upper limbs after stroke. The functional assessment range is an average of 19 sub-items with a range from 0 to 3, with 0 (meaning did not attempt) to 5 (meaning normal). ARAT Day 90 - is a measure of the functional assessment change from baseline to 90 days after 6-months of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jianguo Zhang, MD, Principal Investigator — Department of Neurosurgery, Beijing Tiantan Hospital, Capital Medical University, Beijing, China; Zixiao Li, MD, Principal Investigator — Department of Neurology, Beijing Tiantan Hospital, Capital Medical University, Beijing, China
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No